CLINICAL TRIAL: NCT03596411
Title: Refleeve : A Retrospective Study to Evaluate the Prevalence of the Barett's Esophagus by Gastro-osephagal Endoscopy in Morbid Obese Patients Treated by Sleeve Gastrectomy and the Advantage of the Systematic Detection in the Prevention of Esophageal Carcinoma
Brief Title: The Detection of Barrett's Esophagus by Gastrointestinal Endoscopy Prevents Esophageal Carcinoma in Morbid Obese After Sleeve Gastrectomy
Acronym: Refleeve
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: Cohort 2018
Record Dates: First submitted 2018-05-17; First posted 2018-07-23 (Actual); Last update posted 2018-07-23 (Actual); Status verified 2018-05

CONDITIONS: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Severe Gastroesophageal reflux disease (GERD) leading to a chronic aggression of esophagus mucosa, called Barrett's esophagus is a main complication of Sleeve gastrectomy for morbid obesity. Barrett's esophagus is considered as a early stage of neoplastic transformation to adenocarcinoma. Since this last years, six european bariatric centers have adopted the policy to realize endoscopy before and five years or more after sleeve gastrectomy. Investigators worked out a database comprizing the Endoscopic features and patient characteristics. Refleeve projet aim to analyse the long term follow-up datas of 100 patients, evaluate the prevalence of Barret's esophagus and investigate the advantage of the systemetic detection to prevent esophagus adenocarcinomas.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had had SG with a minimum follow-up of 5 years, without signs of Barrett's esophagus before SG;
* An upper GI endoscopy before the SG;
* An upper GI endoscopy indicating that no Barrett's esophagus was present at the time of the SG;
* An upper GI endoscopy done with the scope of searching for the endoscopic anomalies of the Barrett's esophagus according to the international guidelines for the diagnosis of Barrett's esophagus 9.
* Endoscopic biopsies according to the international guidelines for the diagnosis of Barrett's esophagus 9.

Exclusion Criteria:

* SG as a conversional procedure from another bariatric procedure such as the gastric banding;
* No upper GI endoscopy before the SG
* Barrett's esophagus before the SG;
* A second procedure after the SG such as the conversion to Roux-en-Y gastric bypass or duodenal switch;
* An upper GI endoscopy done not following the international guidelines for the diagnosis of Barrett's esophagus9.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Gastroesophagal reflux disease (GERD) in morbid obese after sleeve gastrectomy
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-05-17 (Actual); Primary Completion 2023-05-17 (Estimated); Study Completion 2023-11-17 (Estimated)

PRIMARY OUTCOMES:
Sleeve gastrectomy | 5 years
  Gastroesophageal endoscopic features before and five years after sleeve gastrectomy

SECONDARY OUTCOMES:
Obesity related comorbidity | 5 years
  obesity related comorbidity before and five years or more after sleeve gastrectomy

CONTACTS AND LOCATIONS:
Overall Officials: IANNELLI Antonio, PhD, Principal Investigator — Chirurgie Digestive, CHU de Nice
Locations (1):
- CHU de Nice, Nice, Alpes Maritimes, France